CLINICAL TRIAL: NCT05713110
Title: A Phase II Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of Tazemetostat in Combination With HMPL-689 in Patients With Relapsed/Refractory Lymphoma
Brief Title: A Study of Tazemetostat in Combination With HMPL-689 in Patients With Relapsed/Refractory Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-TAZ-00CH2
Record Dates: First submitted 2022-12-13; First posted 2023-02-06 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Relapsed/Refractory Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — tazemetostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tazemetostat combined with HMP689 open-label treatment arm (Experimental): Dose Escalation Phase (Phase IIa):
  patients with relapsed or refractory lymphoma who have failed standard treatment and have no standard treatment options
  Dose Expansion Phase (Phase IIb):
  Cohort 1 (DLBCL, FL 3b): Histologically confirmed DLBCL, FL 3b (including primary mediastinal B-cell lymphoma) with relapsed/refractory disease ；
  Cohort 2 (FL) patients with histologically confirmed R/R FL (Grade 1, 2, 3a)；
  Cohort 3 (MCL): Patients with R/R MCL who had prior therapies ；
  Cohort 4 (PTCL): Patients with histologically confirmed R/R PTCL who have failed or cannot tolerate standard therapy
  Interventions: Drug: tazemetostat; Drug: HMPL-689

INTERVENTIONS:
Drug: tazemetostat — Dose Escalation Phase (Phase IIa):
  Tazemetostat (800 mg BID orally) in a therapeutic cycle of 28 days;
  Dose Expansion Phase (Phase IIb):
  Tazemetostat (800 mg BID orally) in a therapeutic cycle of 28 days
Drug: HMPL-689 — Dose Escalation Phase (Phase IIa):
  HMPL-689:20 mg and 30 mg, QD orally in a therapeutic cycle of 28 days.
  Dose Expansion Phase (Phase IIb):
  HMPL-689 (RP2D) in a therapeutic cycle of 28 days

SUMMARY:
A phase II clinical study of tazemetostat combined with HMPL-689 in patients with R/R lymphoma. The study includes 2 phases: dose escalation phase (phase IIa) and expansion phase (phase IIb).

DETAILED DESCRIPTION:
Dose Escalation Phase (Phase IIa ):Including 10-20 patients for dose escalation, the enrollment will continue until about 10 patients in the dose group with response, as to determine Recommended Phase II dose (RP2D).

Dose Expansion Phase (Phase IIb):Multiple expansion cohorts will be set up according to different tumor types, and about 15-20 patients will be enrolled in each cohort to further observe the anti-tumor effect of Tazemetostat combined with HMPL-689 in different pathological types of R/R lymphoma.

This study is expected to enroll 85-140 patients total in Phase IIa and phase IIb.

ELIGIBILITY:
Criteria: Inclusion Criteria:

1. Willing and able to give informed consent, as documented by signed ICF
2. Age ≥ 18 years
3. Patients with histologically confirmed R/R lymphoma:

   • Phase IIa （dose escalation study）: patients with relapsed or refractory lymphoma who have failed standard treatment and have no standard treatment options

   • Phase IIb（ expansion Study ）: Cohort 1 (DLBCL, FL 3b) Histologically confirmed DLBCL, FL 3b (including primary mediastinal B-cell lymphoma) with relapsed/refractory disease

   Cohort 2 (FL) patients with histologically confirmed R/R FL (Grade 1, 2, 3a)

   Cohort 3 (MCL): Patients with R/R MCL who had prior therapies

   Cohort 4 (PTCL): Patients with histologically confirmed R/R PTCL who have failed or cannot tolerate standard therapy
4. Patients must have at least one measurable lesion
5. Life expectancy ≥ 12 weeks
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
7. Adequate bone marrow function, renal function and hepatic function:
8. Currently human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV), or cytomegalovirus (CMV) is inactive
9. Female patients of childbearing potential must agree to use a double contraception method and male patients with partners of childbearing potential must also use an effective double contraception method during the study period and for 3 months after the final dose

Exclusion Criteria:

1. Patients who have previously used EZH2 inhibitors and PI3K inhibitors, or previously could not tolerate EZH2 inhibitors or PI3K inhibitors
2. Patients with brain metastases or leptomeningeal invasion
3. Has thrombocytopenia, neutropenia, or anemia of Grade ≥3 (per CTCAE 5.0 criteria) and any prior history of myeloid malignancies, including myelodysplastic syndrome (MDS / AML/MPN)
4. Has abnormalities known to be associated with MDS (e.g. del 5q, chr 7 abn) and multiple primary neoplasms (MPN) (e.g. JAK2 V617F) observed in cytogenetic testing and DNA sequencing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Dose Escalation Phase (Phase IIa):To evaluate the safety, tolerability, and determine the maximum tolerated dose (MTD) and/or RP2D of Tazemetostat in combination with HMPL-689 in patients with R/R lymphoma | from Cycle 1 Day 1 up to Cycle 1 Day 28 (each cycle is 28 days)
  Occurrence of Dose Limiting Toxicities (DLTs) During the DLT Observation Period
Dose Expansion Phase (Phase IIb):To evaluate the ORR of Tazemetostat in combination with HMPL-689 in patients with lymphoma | from Cycle 1 Day 1 to PFS (each cycle is 28 days)
  Percentage of patients with Complete Response(CR) or Partial Response(PR) as the best response evaluated in accordance with Lugano2014
Dose Expansion Phase (Phase IIb):To evaluate the DCR of Tazemetostat in combination with HMPL-689 in patients with lymphoma | from Cycle 1 Day 1 to PFS (each cycle is 28 days)
  the proportion of patients with CR or PR or stable disease (SD) as the best response with Lugano2014
Dose Expansion Phase (Phase IIb):To evaluate the DOR of Tazemetostat in combination with HMPL-689 in patients with lymphoma | from Cycle 1 Day 1 to PFS (each cycle is 28 days)
  as the time from the first appearance of CR or PR to PD or death for any reason (whichever comes first), in the patients with objective response with Lugano2014)
Dose Expansion Phase (Phase IIb):To evaluate the PFS of Tazemetostat in combination with HMPL-689 in patients with lymphoma | from Cycle 1 Day 1 to PFS (each cycle is 28 days)
  the proportion of patients with CR or PR or stable disease (SD) as the best response with Lugano2014

SECONDARY OUTCOMES:
Dose Escalation Phase (Phase IIa):Objective Response Rate (ORR) | From baseline to final assessment at end of safety follow-up visit(through study completion, an average of 2 years)
  Percentage of patients with Complete Response (CR) or Partial Response (PR) as the best response evaluated in accordance with Lugano 2014
Dose Escalation Phase (Phase IIa)-Complete Response Rate (CR rate) | From baseline to final assessment at end of safety follow-up visit(through study completion, an average of 2 years)
  Percentage of patients with Complete Response (CR) as the best response evaluated in accordance with Lugano 2014
Dose Escalation Phase (Phase IIa)-Disease control rate (DCR) | From baseline to final assessment at end of safety follow-up visit(through study completion, an average of 2 years)
  the proportion of patients with CR or PR or stable disease (SD) as the best response
Dose Escalation Phase (Phase IIa)-Duration of response (DoR) | From baseline to final assessment at end of safety follow-up visit(through study completion, an average of 2 years)
  as the time from the first appearance of CR or PR to PD or death for any reason (whichever comes first), in the patients with objective response
Dose Escalation Phase (Phase IIa)-Time to response (TTR) | From baseline to final assessment at end of safety follow-up visit(through study completion, an average of 2 years)
  the time from the first dose of Tazemetostat in combination with HMPL-689 to the first objective response
Dose Escalation Phase (Phase IIa)-Progression-free survival (PFS) | From baseline to final assessment at end of safety follow-up visit(through study completion, an average of 2 years)
  time from the first dose of study treatment to PD or death for any reason, whichever comes first
Dose Escalation Phase (Phase IIa)-Overall survival (OS) | From baseline to final assessment at end of safety follow-up visit(through study completion, an average of 2 years)
  time from the first dose of study treatment to death for any reason
  time from the first dose of study treatment to death for any reason
Dose Expansion Phase (Phase IIb)-Evaluation of Tazemetostat safety and tolerability in Combination with HMPL-689 in Patients with R/R Lymphoma | From baseline to final assessment at end of safety follow-up visit(through study completion, an average of 2 years)
  Incidence, severity, and causality to study drug of treatment-emergent adverse events (TEAEs) as determined by the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI-CTCAE 5.0)
Geomean maximum concentration (Cmax) of tazemetostat and its metabolite EPZ-6930 in blood | Cycle (C) 1, Day (D) 1: predose of first administration (PoFA); 0.5, 1, 2, 4, 6, 8, and 12 hours postdose. C1D15: PoFA; 0.5, 1, 2, 4, 6, 8, and 12 hours postdose. C1D2, C1D16, C2D1, C3D1 and C4D1: PoFA
  Cmax is defined as the maximum observed concentration that a drug achieves in a test area of the body after the drug has been administered. Plasma concentration-time profiles of tazemetostat and EPZ-6930 will be plotted using non-compartmental analysis and will be analyzed to determine Cmax. Cmax will be summarized as the geomean and geomean CV% for all participants.
Median time to reach maximum concentration (Tmax) of tazemetostat and its metabolite EPZ-6930 in blood | Cycle (C) 1, Day (D) 1: predose of first administration (PoFA); 0.5, 1, 2, 4, 6, 8, and 12 hours postdose. C1D15: PoFA; 0.5, 1, 2, 4, 6, 8, and 12 hours postdose. C1D2, C1D16, C2D1, C3D1 and C4D1: PoFA
  Tmax is defined as the time from dosing to reach the maximum observed concentration a drug achieves in a specified compartment or test area of the body after the drug has been administered. Plasma concentration-time profiles of tazemetostat and EPZ-6930 will be plotted using non-compartmental analysis and will be analyzed to determine Tmax. Tmax will be summarized as the median (min, max) for all participants.
Geomean area under the drug concentration-time curve (AUC) of tazemetostat and its metabolite EPZ-6930 after administration of tazemetostat | Cycle (C) 1, Day (D) 1: PoFA; 0.5, 1, 2, 4, 6, 8, and 12 hours postdose. C1D15: PoFA; 0.5, 1, 2, 4, 6, 8, and 12 hours postdose.
  AUC represents the total drug exposure over a defined period of time. AUC will be calculated using the linear trapezoidal rule. Plasma concentrations of tazemetostat and EPZ-6930 will be analyzed using a non-compartmental analysis approach to determine individual participant estimates of AUC. AUC will be summarized as the geomean and geomean CV% for all participants
Geomean minimum observed concentration at steady-state (Cmin) of tazemetostat and its metabolite EPZ-6930 in blood | C1D15, C1D16, C2D1, C3D1 and C4D1: PoFA
  Cmin is defined as the minimum observed concentration at steady-state during one dosing interval. Cmin will be summarized as the geomean and geomean CV% for all participants.
Geomean maximum concentration (Cmax) of HMPL-689 in blood | Cycle (C) 1, Day (D) 1: predose of first administration (PoFA); 0.5, 1, 2, 4, 6, 8, 12 and 24 (C1D2, PoFA) hours postdose. C1D15: PoFA; 0.5, 1, 2, 4, 6, 8, 12 and 24 (C1D16, PoFA) hours postdose. C2D1, C3D1 and C4D1: PoFA
  Cmax is defined as the maximum observed concentration that a drug achieves in a test area of the body after the drug has been administered. Plasma concentration-time profiles of HMPL-689 will be plotted using non-compartmental analysis and will be analyzed to determine Cmax. Cmax will be summarized as the geomean and geomean CV% for all participants.
Median time to reach maximum concentration (Tmax) of HMPL-689 in blood | Cycle (C) 1, Day (D) 1: predose of first administration (PoFA); 0.5, 1, 2, 4, 6, 8, 12 and 24 (C1D2, PoFA) hours postdose. C1D15: PoFA; 0.5, 1, 2, 4, 6, 8, 12 and 24 (C1D16, PoFA) hours postdose. C2D1, C3D1 and C4D1: PoFA
  Tmax is defined as the time from dosing to reach the maximum observed concentration a drug achieves in a specified compartment or test area of the body after the drug has been administered. Plasma concentration-time profiles of HMPL-689 will be plotted using non-compartmental analysis and will be analyzed to determine Tmax. Tmax will be summarized as the median (min, max) for all participants
Geomean area under the drug concentration-time curve (AUC) of HMPL-689 after administration of HMPL-689 | Cycle (C) 1, Day (D) 1: predose of first administration (PoFA); 0.5, 1, 2, 4, 6, 8, 12 and 24 (C1D2, PoFA) hours postdose. C1D15: PoFA; 0.5, 1, 2, 4, 6, 8, 12 and 24 (C1D16, PoFA) hours postdose
  AUC represents the total drug exposure over a defined period of time. AUC will be calculated using the linear trapezoidal rule. Plasma concentrations of HMPL-689 will be analyzed using a non-compartmental analysis approach to determine individual participant estimates of AUC. AUC will be summarized as the geomean and geomean CV% for all participants.
Geomean minimum observed concentration at steady-state (Cmin) of HMPL-689 in blood | C1D15, C1D16, C2D1, C3D1 and C4D1: PoFA
  Cmin is defined as the minimum observed concentration at steady-state during one dosing interval. Cmin will be summarized as the geomean and geomean CV% for all participants
To investigate the preliminary efficacy and PK correlation | through study completion, an average of 2 years
  The efficacy of participants as assessed by Lugano2014 from different dose groups, to assess the correlation of efficacy and PK of tazemetostat and HMPL-689
To investigate the preliminary tolerability and PK relationship | through study completion, an average of 2 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 from different dose groups, to assess the correlation of safety and PK of tazemetostat and HMPL-689

CONTACTS AND LOCATIONS:
Overall Officials: Bin Yang, Study Director — Hutchison Medipharma Limited
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No